CLINICAL TRIAL: NCT04416386
Title: Does Vitamin C Level Effect Postoperative Analgesia in Orthognathic Surgery: a Preliminary Study?
Brief Title: Vitamin C Level Effect in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Other Study IDs: Medipol Hospital 12
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Maxillofacial Abnormalities; Maxillofacial Injuries; Maxillofacial Trauma
MeSH Terms: conditions — Maxillofacial Abnormalities; Maxillofacial Injuries | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vitamin C — Pre and post-operative blood plasma levels of vitamin C will be investigated

SUMMARY:
Comparing the pre and post-operative blood plasma levels of vitamin C according to oxidative stress and investigate the correlation between post-operative analgesia requirement and vitamin C levels following orthognathic surgery.

DETAILED DESCRIPTION:
Vitamin C (ascorbic acid) is a water-soluble vitamin that has many functions include antioxidant, neuroprotective, neuromodulator and co-factor for various enzymes or chemical reactions. Primarily ascorbic acid is the most potent non-enzymatic antioxidant agent in an extracellular fluid which is crucial for defense against oxidative stress. Recent clinical studies have shown that trauma or surgery may lead to oxidative stress and plasma vitamin C level decreases due to body demand that most likely caused by oxidative stress.

Pain is defined as an unpleasant sensory and emotional experience associated with actual or potential tissue damage. One of the major purposes in the management of post-operative pain is to minimize the dose of medications to reduce side effects while providing adequate analgesia.

In orthopedic surgery and management of postherpetic neuralgia oral vitamin C supplementation significantly reduced pain. However, the decrease in vitamin C concentration,the effects on antinociception and postoperative pain are not fully understood.

In this study, investigators aimed to compare pre and post-operative blood plasma levels of vitamin C after orthognathic surgery and investigate a correlation between post-operative analgesia requirement and vitamin C levels without vitamin C administration.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for orthognatic surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 19 Years to 38 Years | Sex: All
Age Groups: Adult
Study Population: Orthognathic surgery patients aged between 19-38 years (mean age 27.17) with ASA I and ASA II status will be included in this randomized prospective study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Blood plasma levels of vitamin C | Change from baseline blood plasma levels of vitamin C at postoperative 1, 2, 4, 8, 16 hours
  Pre and post-operative blood plasma levels of vitamin C

SECONDARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption levels at postoperative 1, 2, 4, 8, 16 hours
  Postoperative opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Fukushima R, Yamazaki E. Vitamin C requirement in surgical patients. Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):669-76. doi: 10.1097/MCO.0b013e32833e05bc. PMID 20689415
- [Background] Jeon Y, Park JS, Moon S, Yeo J. Effect of Intravenous High Dose Vitamin C on Postoperative Pain and Morphine Use after Laparoscopic Colectomy: A Randomized Controlled Trial. Pain Res Manag. 2016;2016:9147279. doi: 10.1155/2016/9147279. Epub 2016 Oct 30. PMID 27872555
- [Background] Pirbudak L, Balat O, Cekmen M, Ugur MG, Aygun S, Oner U. Effect of ascorbic acid on surgical stress response in gynecologic surgery. Int J Clin Pract. 2004 Oct;58(10):928-31. doi: 10.1111/j.1742-1241.2004.00022.x. PMID 15587771